CLINICAL TRIAL: NCT03498391
Title: A Study of Human Multi-Sensory Integration: A Neurophysiologic Correlate of Conscious Perception
Brief Title: A Study of Human Multi-Sensory Integration
Acronym: MSI
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the impact of COVID-19
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 829800
Record Dates: First submitted 2018-03-12; First posted 2018-04-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia Awareness
MeSH Terms: conditions — Intraoperative Awareness | interventions — Propofol; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Propofol (Experimental): Propofol sedation titrated to clinical effect as measured by Richmond Agitation-Sedation Scale.
  Interventions: Drug: Propofol
- Ketamine (Experimental): Ketamine sedation titrated to clinical effect as measured by Richmond Agitation-Sedation Scale.
  Interventions: Drug: Ketamine Injectable Product

INTERVENTIONS:
Drug: Propofol — Titration of propofol to minimal and moderate sedation as measured by Richmond Agitation-Sedation Scale with behavioral task performance over several hours.
  Other Names: Diprivan
  Arms: Propofol
Drug: Ketamine Injectable Product — Titration of ketamine to minimal and moderate sedation as measured by Richmond Agitation-Sedation Scale with behavioral task performance over several hours.
  Other Names: Ketalar
  Arms: Ketamine

SUMMARY:
The primary aim of this study is to determine whether spatiotemporal characteristics of multisensory evoked potentials can be used as a marker of consciousness (awareness) under anesthesia.

The secondary aim is to characterize changes in the characteristics of evoked potentials under anesthesia in both single sensory modality (visual, auditory) and across sensory modalities.

DETAILED DESCRIPTION:
This is a prospective, dual parallel arm human subject study aimed at determining the relationship between level of sedation (consciousness) and features of multi and uni-sensory evoked potentials with the ultimate goal of developing novel means of detecting consciousness under anesthesia with potential for application to other clinical settings such as brain injury. For this purpose, the investigators have chosen two anesthetics with fundamentally distinct mechanisms of action: propofol and ketamine.

The study will involve healthy compensated volunteers. On the day of the study, an EEG cap will be applied to the participant for monitoring brain activity and an intravenous line will be placed for drug administration. Blood pressure, ECG, pulse oxymetry, and end-tidal carbon dioxide (from nasal cannula) will be monitored. Supplemental oxygen will be administered using a nasal cannula. Subjects will then perform the behavioral tasks in the awake state for approximately 1 hour.

After this phase is complete, participants will receive either propofol or ketamine (chosen permuted block randomization) using a clinician bolus/infusion strategy titrated to Richmond Agitation-Sedation Scale score of -1 (see above). Once the desired sedation level is achieved, subjects will once again complete the behavioral tasks. After the completion of this phase (approximately 1 hour) the anesthetic dose will be increased to attain Richmond Agitation-Sedation Scale -3 to -4. At this level of sedation subjects will not be able to do the behavioral task and only the evoked potentials will be recorded. Upon completion of this phase (approximately 1 hour), sedation level will be decreased to return the subject to a Richmond Agitation-Sedation Scale of -1 and once again the tasks will be repeated.

Finally, the anesthetic infusion will be stopped. Once the Richmond Agitation-Sedation Scale score of 0 is attained, participants will once again perform the behavioral task (approximately 1 hour). This will conclude the experimental phase of the trial. Subjects will be monitored until clinically established discharge criteria are met. This includes adequate respiration, blood pressure, oxygen saturation and activity level. No formal follow-up is required; however, subjects will be called 24 hours after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ages 18-65 years old
* American Society of Anesthesiologists (ASA) Physical Status I or II (i.e. healthy)
* Body Mass Index <30 kg/m2
* Easily visible uvula

Exclusion Criteria:

* Contraindications to administration of either propofol or ketamine
* Allergy to either one of the medications or preservative in which it is diluted.
* History (or current) seizure disorder
* Contraindications to anesthesia
* Significant cardiovascular disease (e.g. h/o hypertension, arrhythmias, myocardial infarction, congestive heart failure, congenital heart defects, coronary artery disease)
* Increased risk factors for difficult intubation and/or ventilation
* Obesity (BMI>=30 kg/m2)
* Mallampati class > 2.
* History of or current obstructive sleep apnea.
* Increased risk of aspiration
* Any per oral intake within 8 hours of anesthetic exposure
* Conditions that delay gastric emptying (e.g. obesity, hiatal hernia, gastro esophageal reflux disease, pregnancy, etc.)
* Pulmonary disease (e.g. chronic obstructive pulmonary disorder, asthma requiring rescue inhaler within last month, emphysema, pulmonary hypertension, pulmonary fibrosis etc).

  * Neurological disease. Patients with history of strokes, seizures, brain surgery, brain tumor, increased intracranial pressure.
  * Psychiatric disease. History of or presents of psychosis, schizophrenia, schizo-affective disorder.
  * Specific Medication Current Use. History of or current intake of antipsychotics or sedatives.
  * Drug abuse. History of or current use of illegal drugs such as stimulants or depressants.
  * Pregnancy or breastfeeding
  * Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Multi-sensory Evoked Responses Measured using Electroencephalography | 2-6 hours per subject
  The primary study endpoint is multi-sensory evoked responses measured using EEG in units of millivolts squared per hertz at Richmond Agitation and Sedation Scale scores of 0, -1, -2, -3 and -4. Multisensory evoked responses will be compared to those evoked by each uni-sensory modality (auditory and visual) individually. Evoked responses will be assessed in the frequency domain using spectral analysis techniques which quantify power of each neuronal oscillation (e.g. alpha, delta, theta and gamma) in terms of mV^2/Hz. Analysis will be performed separately during the period before drug administration and at different levels of sedation quantified with RASS scores. The investigators will test the hypothesis that with increasing doses of intravenous anesthetics, audiovisual (multisensory) responses will approximate algebraic sum of neuronal responses elicited by visual and auditory stimuli presented separately.

SECONDARY OUTCOMES:
Single Modality Evoked Potentials | 2-6 hours per subject
  The secondary endpoint is to use EEG recordings to demonstrate changes in the characteristics of evoked potentials under anesthesia using single sensory modality (visual, auditory) and across sensory modalities. Conventional evoked potentials will be computed as average waveforms aligned with respect to stimulus onset on a channel-by-channel basis.

CONTACTS AND LOCATIONS:
Overall Officials: Max Kelz, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Perelman School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No